CLINICAL TRIAL: NCT07127055
Title: Modulation of Metabolic Parameters Among Obese Diabetic Individuals Through a Gluten-Free Diet
Brief Title: Gluten Free Diet on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sana Noreen, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UOL/IREB/25/09/0008
Record Dates: First submitted 2025-08-08; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Syndrome; Lipid Profile; HOMA-IR; Weight Change, Body
MeSH Terms: conditions — Metabolic Syndrome; Body Weight Changes | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (T1): Conventional treatment + Standard Diet (Placebo Comparator): Group T1 received a standard diet, 1800 kcal/day for 12 weeks
  Interventions: Other: No intervention
- Treatment Group T2: Conventional treatment + Gluten-free diet 1800 Kcal/day (Experimental): Group T2 received a gluten-free diet for 12 weeks
  Interventions: Other: gluten free diet

INTERVENTIONS:
Other: No intervention — Control group will take standard diet
  Arms: Control group (T1): Conventional treatment + Standard Diet
Other: gluten free diet — This group received gluten free diet
  Arms: Treatment Group T2: Conventional treatment + Gluten-free diet 1800 Kcal/day

SUMMARY:
This study benefits the community by highlighting the potential of a gluten-free diet as a non-pharmacological, effective approach to managing obesity and type 2 diabetes. By demonstrating significant improvements in weight, blood sugar, lipid levels, and liver function, it supports dietary modification as a practical approach to enhancing metabolic health. The findings can inform public health initiatives, raise community awareness about the role of nutrition in disease management, and promote personalized dietary interventions, ultimately contributing to better prevention and control of chronic metabolic conditions.

DETAILED DESCRIPTION:
2.1. The study received ethical approval from the Institute Research Ethics Board (IREB), University of Lahore (UOL/IREB/25/09/0008). Informed consent was obtained from all participants, who were fully briefed on the study's purpose, procedures, risks, and benefits, with the option to ask questions and withdraw at any time.

2.2. Study design The research trial, a randomized controlled trial (RCT), was carried out at the Dilawar Hussain Foundation, Diabetes Management Center, Lahore, Pakistan.

An intervention with a tailored gluten-free diet of 1800 kcal/day was planned. 2.3. Methods of data collection A total of 115 volunteers who met the inclusion criteria were recruited into the study. Seven participants left the study due to personal issues; a total of 108 patients left, which were divided into two equal groups (n=54 in each group).

Participants were randomly allocated to two study groups. Group T1 received a standard diet, whereas Group T2 received a gluten-free diet for 12 weeks. An 1800 kcal/day diet was nutritionally comparable, 50-55% of calories were from carbohydrates, 15-20% protein, and 25-30% fat. Fiber in the form of fruits, vegetables, legumes, and the right grains. The gluten-free variant omitted all sources of wheat, rye, and barley and thus was the ideal option for those needing a gluten-free diet. Follow-up sessions on alternate days were used to guarantee compliance throughout the intervention period, where dietary adherence was checked and reinforced. At the end of week 12th, biochemical tests were performed for all the subjects. The post-interventional measurements between the two groups were then compared to assess the metabolic effects of the gluten-free diet. This comparison was used to test the main hypothesis of the study.

2.4. Parameters for assessment The final dataset comprised anthropometric data: weight, height, body mass index (BMI), and waist circumference, 24-hour dietary recall, as outlined. In addition, fasting glucose level, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), systolic and diastolic blood pressure, and lipid profiles in serum (LDL, HDL, and total cholesterol) were measured using the same procedure.

2.5 Statistical analysis Data analysis was performed using SPSS version 25. Continuous variables were summarized as mean ± standard deviation, while categorical variables were presented as frequencies and percentages. Baseline and post-study comparisons were made using paired sample t-tests, with significance set at p ≤ 0.05 .

ELIGIBILITY:
Inclusion Criteria:

* Patients who were obese diabetic adults of both genders, aged 30 to 55 years,
* body mass index (BMI) > 25 kg/m²,
* fasting glucose level > 135 mg/dL,
* elevated parameters of lipid profile,
* blood pressure > 135/85 mmHg,
* Insulin Resistance (HOMA-IR) > 2.57

Exclusion Criteria:

* Patients with a diagnosis of celiac disease,
* irritable bowel syndrome,
* some cancers,
* genetic illnesses,
* respiratory illnesses, and psychiatric illnesses

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurement | 12 weeks
  Baseline anthropometric measurements, including weight, height, BMI, and waist circumference, were recorded following standard clinical procedures. Weight was measured with a calibrated electronic scale while subjects wore light clothing and were barefoot. Height was measured using a calibrated stadiometer with subjects standing erect and barefoot. BMI was calculated as weight (kg) divided by height squared (m²). Waist circumference was measured with a non-elastic tape placed midway between the lowest rib and iliac crest, ensuring the tape touched the skin without compressing it.
24-hour dietary recall method | 12 WEEKS
  The 24-hour dietary recall method was used to assess participants' intake through structured interviews. A multi-pass approach ensured detailed and accurate reporting of food, portion sizes, and preparation methods. Recalls on non-consecutive days captured dietary variation, and data were analyzed using validated tools to estimate nutrient intake.
Assessment of Lipid Profile (mg/dL) | 12 Weeks
  Blood samples for baseline and follow-up tests were collected in EDTA-treated tubes to assess hematological parameters. Total cholesterol (TC), triglycerides (TG), and HDL levels were measured using an enzymatic colorimetric method, whereas LDL-C concentration was checked with the help of a formula. The following equation was used to calculate very low-density lipoprotein cholesterol (VLDL).
  VLDL - c (mg∕dL) = TG∕5 LDL = Total cholesterol - (HDL + VLDL)

SECONDARY OUTCOMES:
Assessment of liver function (U/L) | 12 Weeks
  Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine aminotransferase (ALT) were estimated.
HOMA-IR | 12 Weeks
  HOMA-IR was calculated to estimate insulin resistance from fasting blood glucose and fasting insulin. Blood was obtained from the subjects after an overnight fast of 8-12 hours. Serum insulin was measured by a validated enzyme-linked immunosorbent assay (ELISA), and fasting blood glucose was measured by a glucose oxidase assay. HOMA-IR value was subsequently calculated by the following formula:
  HOMA-IR = Fasting Insulin (µU/mL)×Fasting Glucose (mg/dL)/405 This method provides an approximation of insulin resistance, with higher values being related to higher resistance. A HOMA-IR above 2.57 was used to denote insulin resistance in the present study

CONTACTS AND LOCATIONS:
Locations (1):
- Sana Noreen, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data will be accessible upon submission. Access will be provided through a secure data-sharing platform. Supporting documents, including the study protocol and statistical analysis plan, will also be available.
Supporting Information: Study Protocol

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30362336/